CLINICAL TRIAL: NCT00486460
Title: Phase III Trial of Gemcitabine, Curcumin and Celebrex in Patients With Advance or Inoperable Pancreatic Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: TASMC-07-NA-132-CTIL
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Last update posted 2007-06-14 (Estimated); Status verified 2007-06

CONDITIONS: Pancreatic Cancer
Keywords: Locally advanced or metastatic adenocarcinoma of the; pancreas; confirmed by histology or cytology; Inoperatable
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Curcumin; Celecoxib

INTERVENTIONS:
Drug: Gemcitabine
Drug: Curcumin
Drug: Celebrex

SUMMARY:
Pancreatic cancer is an aggressive disease with an extremely poor prognosis. It is the forth leading cause of cancer-related fatalities, with an estimated one-year and five-year survival rate of 21% and 5%, respectively. Despite recent progress, the median survival time is 6-10 months for patients with locally advanced disease and 3-6 months for metastatic disease (1). The anti-metabolite gemcitabine has become the standard chemotherapy for locally advanced and metastatic pancreatic cancer, after demonstrating an improved rate of clinical benefit response and an overall survival advantage over 5-FU (2). In addition to its clinical effectiveness gemcitabine has a manageable toxicity profile, making it an attractive agent to investigate in combination with newer agents. Series of phase III trials were conducted examining the efficacy of the combination of gemcitabine and a second cytotoxic agent, including 5-FU, cisplatin, oxaliplatin and irinotecan. These gemcitabine doublets demonstrated no survival advantage over single-agent gemcitabine (3-6). However, the rationale for continuing to study gemcitabine-based combinations remains compelling.

Curcumin (diferuloylmethane) is a natural compound derived from the rhizome of Curcuma Longa, an East Indian plant, commonly called turmeric. It has been shown to possess potent anti-inflammatory and anti-oxidative properties, for which it has a long history of dietary use as a food additive. Curcumin has also a potent anti-proliferative effects against a variety of cancer cell lines in vitro, which stem from its ability to modulate many intracellular signal transduction pathways (7). Human phase I-II studies found curcumin to be safe, and indicated no dose-limiting toxicity when taken by mouth at doses up to 10 g/day (8, 9). This data, together with the dismal therapeutic options available for pancreatic cancer patients, suggest that curcumin warrants investigation in this setting. Investigators from MD Anderson Cancer Center and Rambam Medical Center in Haifa, have recently initiated, separately, a phase II study of single agent Curcumin in patients with pancreatic cancer (10).

One of the lessons learned from cancer research in recent decades is that combination strategies can provide dramatic improvement in a therapy's safety and efficacy over mono-therapeutic regiments, especially if the combined drugs differ in their mode of action. In a recent paper that was accepted for publication we demonstrated, in vitro, the mechanism, clinical importance and implications of a novel combinatorial therapy, of celecoxib and curcumin, that was discovered in our lab, in inhibiting the growth of several pancreatic cell lines. P-34 (expressing high levels of COX -2), MiaPaca (Expressing low levels of COX-2) and Panc-1 (no expression of COX -2) cell lines were exposed to different concentrations of celecoxib (0-40µM), curcumin (0-20µM) and their combination. In P-34 cells, curcumin synergistically potentiated the inhibitory effect of celecoxib on cell growth. The growth inhibition was associated with inhibition of proliferation and induction of apoptosis.

These experiments further demonstrate, for the first time, that the combination effect is correlated with synergistic augmentation of apoptosis and involves down-regulation of COX-2 protein.

The present study evaluates gemcitabine in combination with curcumin and celecoxib for patients with pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic adenocarcinoma of the pancreas, confirmed by histology or cytology.
* No prior chemotherapy for pancreatic cancer.
* Performance status 0-2 (ECOG scale).
* Age ≥ 18 y.
* Adequate hematologic function (ANC ≥ 1500/mm³, platelet count ≥ 100,000/mm³).
* Adequate hepatic function (total bilirubin ≤ 2.0xUNL and AST, ALT and AP ≤ 5.0xUNL)
* Adequate renal function (creatinine ≤ 2.0).
* Signed informed consent.

Exclusion Criteria:

* A history of treated or active central nervous system involvement by the tumor or active neurological disease.
* Prior radiation. Patients with disease outside the irradiation field or documented disease progression of previously irradiated disease are eligible.
* Unstable medical condition, including uncontrolled diabetes mellitus or hypertension, active infection, unstable CHF, uncontrolled arrhythmias or unstable coagulation disorders.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Arber Nadir, M.D, Msc, MHA, Principal Investigator — University of Tel Aviv
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel